CLINICAL TRIAL: NCT02895529
Title: A Multicenter, Randomized Trial Comparing The Efficacy of Intravenous Followed by Oral Itraconazole With Intravenous Caspofungin For Empiric Antifungal Therapy in Neutropenic Subjects With Hematological Malignancy
Brief Title: A Study Comparing the Efficacy of Intravenous Followed by Oral Itraconazole With Intravenous Caspofungin For Empiric Antifungal Therapy in Neutropenic Participants With Hematological Malignancy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study is a commitment for license renew, we target on Apr19 submission, considering timeline, a cut off should be scheduled in Apr18.
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108202; R051211FUN4057 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Itraconazole; Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itraconazole (Experimental)
  Interventions: Drug: Itraconazole
- Caspofungin (Active Comparator)
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Itraconazole — Participants will receive 200 milligram (mg) of itraconazole intravenously (IV) twice daily on Day 1 and Day 2, followed by 200 mg once daily through Day 14. From Day 15 to Day 28, participants will receive 200 mg (20 milliliters [mL]) of itraconazole oral solution orally twice daily. Participants, who are not suitable for oral administration of itraconazole based on the investigator's judgment, will receive 200 mg of itaconazole IV once daily from Day 15 to Day 28.
  Arms: Itraconazole
Drug: Caspofungin — Participants will receive 70 mg of caspofungin IV once daily on Day 1 followed by 50 mg IV infusion once daily thereafter through Day 28.
  Arms: Caspofungin

SUMMARY:
The purpose of this study is to investigate the hypothesis that the efficacy of intravenous (IV) itraconazole followed by oral itraconazole is non-inferior to that of intravenous caspofungin as empiric therapy for suspected fungal infection participants with fever and neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be hospitalized with hematologic malignancy treated by myelosuppressive therapy and/or Hematopoietic stem cell transplantation
* Participant must have a diagnosis of neutropenia with neutrophil count < 500/microliters (mcL) (0.5 × 10^9/ liters [L]) for at least 96 hours at screening
* Participant must have a diagnosis of fever and meet the following criteria: 1) Oral/rectal temperature greater than or equal to (>=) 38 degree celsius or axillary temperature (>=) 37.5 degree celsius and is not considered related to blood products transfusion or drug fever, 2) Not responding to broad-spectrum gram-positive and gram-negative antibiotics for 4-7 days with or without signs and symptoms that potentially attributable to deep fungal infection and 3) Defervescence within 3 days after the first broad-spectrum antibiotics but recurrence afterwards.
* A woman of childbearing potential must have a negative serum (beta human chorionic gonadotropin [b hCG]) and pregnancy test at screening
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study period and until the menstrual period following the end of study treatment

Exclusion Criteria:

* Is concomitantly using other systematic antifungal drugs as empirical treatment
* Has evidence of inadequately managed bacterial infection
* Is currently receiving any Cytochrome P450 3A4 (CYP3A4)-metabolized/P-glycoprotein-transported drugs (including but not limited to cisapride, pimozide, quinidine, dofetilide, levacetylmethadol, terfenadine, astemizole, mizolastine, bepridil, sertindole, 3-hydroxy-3-methyl-glutaryl-coenzyme A reductase (HMG-CoA reductase) inhibitor [for example, simvastatin, lovastatin], oral midazolam, triazolam, ergot alkaloids [eg, dihydroergotamine, ergonovine, ergotamine, methylergonovine] and nisoldipine) that should be prohibited in this study
* Has known allergy, intolerance or hypersensitivity to azole and echinocandin antifungals or its excipients
* Has a contraindication to the use of sodium chloride injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Response Rate Measured by the Percentage of Participants That Achieve all of the Following 5 Composite Endpoints | Up to 36 days
  Response rate in each of the 2 treatment groups will be measured by the percentage of participants that achieve all of the following 5 composite endpoints: 1) survival for 7 days after completion of treatment, 2) absence of breakthrough invasive fungal infection during the study drug administration and within the first 7 days after completion of treatment, 3) successful treatment of baseline fungal infection, 4) defervescence and 5) no premature withdrawal from the study due to drug-related toxicity or lack of efficacy.

SECONDARY OUTCOMES:
Percentage of Participants With Survival for 7 Days After Completion of Treatment | Up to 36 days
Percentage of Participants With Absence of Breakthrough Invasive Fungal Infection | Day 3 up to Day 28 (End of treatment [EoT]) and within 7 days after EoT (Day 29 up to Day 35)
  Absence of breakthrough invasive fungal infection is defined as the clinically or/and microbiologically documented fungal infection with an onset on or after day 3 of the study treatment during the study drug administration and within the first 7 days after completion of treatment.
Percentage of Participants With Successful Treatment of Baseline Fungal Infection | Screening up to Day 3
  Successful treatment of baseline fungal infection is defined as the clinically and microbiologically documented fungal infection with an onset within screening to 2 days after the study treatment.
Percentage of Participants With Defervescence During the Period of Neutropenia | Up to 36 days
  Defervescence is defined as oral/rectal temperature less than (<) 38 degree celsius or axillary temperature (<) 37.5 degree celsius for over 48 hours) during the period of neutropenia.
Percentage of Participants With No Premature Withdrawal From the Study due to Drug-related Toxicity or Lack of Efficacy | Up to 36 days
Response Rate Measured by the Percentage of Participants That Achieve all of the Following 5 Composite Endpoints With Oral Administration of Itraconazole | Up to 36 days
  Response rate will be measured by the percentage of participants (who received oral administration of itraconazole) that achieve all of the following 5 composite endpoints: 1) survival for 7 days after completion of treatment, 2) absence of breakthrough invasive fungal infection during the study drug administration and within the first 7 days after completion of treatment, 3) successful treatment of baseline fungal infection, 4) defervescence and 5) no premature withdrawal from the study due to drug-related toxicity or lack of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (12):
- China (12):
  - Beijign
  - Beijing
  - Changchun
  - Changzhou
  - Fuzhou
  - Guangzhou
  - Guiyang
  - Hefei
  - Shanghai
  - Suzhou
  - Tianjin
  - Zhengzhou

REFERENCES:
- See also: A Multicenter, Randomized Trial Comparing The Efficacy of Intravenous Followed by Oral Itraconazole With Intravenous Caspofungin For Empiric Antifungal Therapy in Neutropenic Subjects With Hematological Malignancy — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108202&attachmentIdentifier=0de79b23-8b15-44f4-88da-5508c86ad8b0&fileName=CR108202_CSR.pdf&versionIdentifier=